CLINICAL TRIAL: NCT02290015
Title: Effectiveness of Acupuncture as a Treatment for Tinnitus: a Randomized Controlled Trial Using 99mTc-ECD SPECT
Brief Title: Acupuncture as a Treatment for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Maura Regina Laureano, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAPESP-2010/14804-6
Record Dates: First submitted 2014-10-28; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Tinnitus
Keywords: Single Photon Emission Computed Tomography; Acupuncture
MeSH Terms: conditions — Tinnitus | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- true acupuncture (Experimental): 12 sessions of ACP treatment were performed twice a week. Before ACP was performed, patients were examined based on the diagnostic pattern of TCM. Then, the appropriate acupoints for treatment were selected according to the tinnitus-related syndrome. The experimental group was treated with true ACP (stimulating selected meridian points), and the control group was treated with sham-ACP (stimulating false meridian points). The patients were blinded to the identity of their treatment group. Disposable stainless steel ACP needles (0.25 x 30 mm, Dong Bang Acupuncture, Korea) were used in both groups. Needles were inserted manually at each meridian point, and the retention time was twenty minutes.
  Interventions: Other: Acupuncture
- sham acupuncture (Sham Comparator): The control group was treated with sham-ACP (stimulating false meridian points). Disposable stainless steel ACP needles (0.25 x 30 mm, Dong Bang Acupuncture, Korea) were used. Needles were inserted manually at each false meridian point, and the retention time was twenty minutes.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — All treatments were performed by the same acupuncturist, who is a medical doctor with more than eight years of clinical and research experience in ACP for tinnitus. Acupoints described as being effective for tinnitus were selected according to TCM theory. Basic points that are manipulated in ACP include GV 20 (Baihui), TE 17 (Yifeng), GB 8 (Shuaigu), SI 19 (Tinggong), GB 2 (Tinghui), TE 21 (Ermen), VC 23 (Lianquan), GB 20 (Fengchi), TE 2 (Yemen), TE 5 (Waiguan), SI 2 (Qiangu), GB 43 (Xiaxi) and GB 41 (Zulinqi). However, several secondary (accessory) acupoints were also added according to TCM and the etiological diagnosis of tinnitus: GV 4 (Mingmen), KI 3 (Taixi), BL 23 (Shenshu), BL 19 (Danshu), BL 18 (Ganshu) and CV 4 (Guanyuan).

SUMMARY:
This trial was a randomized, single-blinded, sham-controlled study, in which the patients were blinded to treatment assignment. First, all candidates underwent audiological testing of hearing thresholds, tympanometry and stapedius reflex tests. The patients who were selected for the study were interviewed to assess and evaluate their condition and then underwent a detailed physical examination that included a complete otorhinolaryngologic examination and a complete blood test. Then, the subjects were randomized to undergo true or sham ACP. Seven days before (baseline) and seven days after twelve acupuncture (ACP) sessions (up to six weeks), which were performed twice a week, all participants underwent 99mTc-ECD SPECT scanning and completed the Portuguese version of the Tinnitus Handicap Inventory (THI), the Visual Analogue Scale (VAS), Hamilton Anxiety Scale (HAS) and the Beck Depression Inventory (BDI). The purpose of this study was to integrate the neuroscience research findings with the clinical research on tinnitus. Thus, a randomized, single-blinded, placebo-controlled trial was implemented to investigate the effect of ACP as a treatment for tinnitus using ethylcysteine dimer single-photon emission computer tomography (99mTc-ECD SPECT).

DETAILED DESCRIPTION:
Acupuncture (ACP) is frequently used to treat tinnitus, the condition defined as the perception of sound in the absence of an external auditory stimulus. However, no information is available regarding the consequences of ACP on the neural architecture and functionality of the brain in tinnitus patients. The aim of this study was to investigate changes in brain activity using ethylcysteine dimer single-photon emission computer tomography (99mTc-ECD SPECT) in patients with tinnitus and normal hearing who underwent ACP treatment. Methods and Findings: This was a randomized, single-blinded, sham-controlled study. The participants were adults (18-60 years old) with either normal hearing or chronic, idiopathic and continuous (+ 3 months) tinnitus. Fifty-seven (57) subjects were randomized to receive true (n=30) or sham (n=27) ACP, and 99mTc-ECD SPECT exams were performed seven days before (baseline) and seven days after twelve ACP sessions (up to six weeks), which were performed twice a week. Secondary outcomes included changes in the Tinnitus Handicap Inventory (THI), the Visual Analog Scale (VAS), the Hamilton Anxiety Scale (HAS) and the Beck Depression Inventory (BDI). Data regarding imaging outcomes were analyzed with Statistical Parametric Mapping (SPM8) software using a factorial design. For secondary outcomes, regression models were built considering two different analytical paradigms: intention-to-treat (ITT; where multiple imputations were conducted due to loss to follow-up) and complete cases. No significant differences in brain perfusion were observed between patients who underwent true versus sham ACP treatment. However, a significant improvement in THI scores at the end of true ACP treatment was observed for all domains (all p < 0.001), with the exception of the catastrophic field. For the other outcome measurements (VAS, BDI and HAS), no significant differences were observed between groups. The small sample size represents a potential limitation of this study. Conclusions: These findings suggest that ACP may improve the impact of tinnitus on daily life, although additional studies are needed to verify the consequences of ACP on the neural architecture and functionality of the brain in tinnitus patients.

ELIGIBILITY:
Inclusion Criteria:

Patients who met all the following conditions were considered for inclusion:

* 18 to 60 years of age
* Existence of typical conditions of subjective and continuous tinnitus, either unilateral or bilateral, for more than three months
* Normal hearing sensitivity in the conventional audiometric range (up to 25 dB from 250 to 8000 Hz) bilaterally and normal immittance measures (type A curve) in both ears

Exclusion Criteria:

The exclusion criteria were as follows:

* Objective, acute or intermittent tinnitus
* History of Ménière's disease
* Tinnitus induced by cerebellopontine angle tumors, cardiovascular disease, or a serious medical or mental illness
* History of central nervous system disease
* Current pregnancy or breast-feeding
* Patients with a lack of willingness or availability to cooperate were also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Ethylcysteinate dimer single-photon emission computer tomography (99mTc-ECD SPECT) | SPECT exam was performed seven days before (baseline) and seven days after acupuncture treatment (up to six weeks)

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | The scale was performed seven days before (baseline) and seven days after acupuncture treatment (up to six weeks)
Visual Analog Scale (VAS) | The scale was performed seven days before (baseline) and seven days after acupuncture treatment (up to six weeks)
Hamilton Anxiety Scale (HAS) | The scale was performed seven days before (baseline) and seven days after acupuncture treatment (up to six weeks)
Beck Depression Inventory (BDI) | The scale was performed seven days before (baseline) and seven days after acupuncture treatment (up to six weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea P Jackowski, PhD, Study Director — Federal University of São Paulo UNIFESP